CLINICAL TRIAL: NCT00238732
Title: A Double-Blind, Randomized, Placebo-and Active-Controlled Efficacy and Safety Study of Bazedoxifene/Conjugated Estrogens Combinations for Treatment of Moderate to Severe Vulvar/Vaginal Atrophy in Postmenopausal Women
Brief Title: Study Evaluating Bazedoxifene/Conjugated Estrogen Combinations in Vasomotor Symptoms Associated With Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3115A1-306
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Vaginal Atrophy
Keywords: Vaginal Atrophy; Postmenopause
MeSH Terms: interventions — bazedoxifene; Estrogens, Conjugated (USP)

INTERVENTIONS:
Drug: Bazedoxifene/Conjugated Estrogen

SUMMARY:
The purpose of this study is to determine whether Bazedoxifine/conjugated estrogens are effective in the treatment of vaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women, aged 40 to 65 years
* Intact uterus
* At least 1 moderate to severe vulvar/vaginal symptom that is most bothersome

Exclusion Criteria:

* Hypersensitivity to estrogens, endometrial hyperplasia, known or suspected estrogen-dependent neoplasia
* Thrombophlebitis, thrombosis or thromboembolic disorders
* Neuro-ocular disease

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2005-10; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Superficial cells (by cervical/vaginal cytologic smear) at screening, and weeks 4 and 12.
Parabasal cells (by cervical/vaginal cytologic smear) at screening, and weeks 4 and 12.

SECONDARY OUTCOMES:
Vaginal pH at screening, and weeks 4 and 12.
Most bothersome moderate or severe vulvar/vaginal atrophy sympton at screening, and weeks 4 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (63):
- United States (63):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Oakland, California
  - San Diego, California
  - Upland, California
  - Denver, Colorado
  - Avon, Connecticut
  - Groton, Connecticut
  - Waterbury, Connecticut
  - Aventura, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Palm Harbor, Florida
  - Palm Springs, Florida
  - Pinnellas Park, Florida
  - Stuart, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Conyers, Georgia
  - Douglasville, Georgia
  - Savannah, Georgia
  - Idaho Falls, Idaho
  - Champaign, Illinois
  - Chicago, Illinois
  - Kansas City, Kansas
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Booklyn Center, Minnesota
  - Chaska, Minnesota
  - Jackson, Mississippi
  - Kansas, Mississippi
  - Creve Cour, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Livingston, New Jersey
  - New Brunswick, New Jersey
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Jamestown, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Erie, Pennsylvania
  - Media, Pennsylvania
  - West Reading, Pennsylvania
  - Hilton Head Island, South Carolina
  - Sioux Falls, South Dakota
  - Nashville, Tennessee
  - Dallas, Texas
  - Denton, Texas
  - Galveston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington

REFERENCES:
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252
- [Derived] Pinkerton JV, Bushmakin AG, Komm BS, Abraham L. Relationship between changes in vulvar-vaginal atrophy and changes in sexual functioning. Maturitas. 2017 Jun;100:57-63. doi: 10.1016/j.maturitas.2017.03.315. Epub 2017 Mar 22. PMID 28539177